CLINICAL TRIAL: NCT06201572
Title: The Value of Smartphone-based Optical Blood Spectrum Imaging (TOI) in Evaluating Renal Function Damage in Hypertensive Emergency Patients
Brief Title: The Value of TOI in Evaluating Renal Function Damage in Hypertensive Emergency Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Hangzhou Normal University (Other)
Responsible Party: Sponsor
Other Study IDs: AH-2023-001
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-11

CONDITIONS: Hypertensive Emergency
MeSH Terms: conditions — Hypertensive Crisis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Observation group
  Interventions: Other: The relationship between TOI composite index and renal function in hypertensive emergency patients was compared
- Control group
- Positive control group

INTERVENTIONS:
Other: The relationship between TOI composite index and renal function in hypertensive emergency patients was compared — The relationship between TOI composite index and renal function in hypertensive emergency patients was compared. The data management platform provides intelligent management of patients' out-of-hospital follow-up, and the dynamic physiological indicators and psychological assessment data of patients are mastered through the hospital port, so as to provide telemedicine guidance for patients, so as to improve the prognosis of hypertensive emergency patients.
  Groups: Observation group

SUMMARY:
TOI was used to measure heart rate, respiration, blood pressure, heart rate variability and psychological stress. At the same time, the patient's urine protein, creatinine, urea nitrogen and other indicators were detected. According to different renal function, they were divided into observation group and control group, and 100 general inpatients with renal insufficiency were selected as positive control group. The relationship between TOI composite index and renal function in hypertensive emergency patients was compared.

DETAILED DESCRIPTION:
TOI technique was used to measure the heart rate, respiration, blood pressure, heart rate variability, psychological pressure, etc. At the same time, the urine protein, creatinine, urea nitrogen and other results of these patients were measured. According to the different renal function, they were divided into observation group and control group, and 100 ordinary hospitalized patients with renal insufficiency were selected as positive control group. The relationship between TOI composite index and renal function in hypertensive emergency patients was compared. The data management platform provides intelligent management of patients' out-of-hospital follow-up, and the dynamic physiological indicators and psychological assessment data of patients are mastered through the hospital port, so as to provide telemedicine guidance for patients, so as to improve the prognosis of hypertensive emergency patients.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure (SBP)>180mmHg
* Diastolic blood pressure (DBP)>120mmHg

Exclusion Criteria:

* Severe head and facial skin injury
* Cerebral hemorrhage or severe shock after admission
* Patients who insist on refusing to participate in this clinical tria
* Patients who could not participate in the study for other reasons.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for acute hypertension from January 2022 to December 2024 with onset time <48 hours and blood pressure measured by standard sphygmomanometer: Systolic blood pressure (SBP)>180mmHg and/or diastolic blood pressure (DBP)>120mmHg, age >18 years old, gender, stable vital signs, good compliance, complete and reliable medical records.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
blood pressure | 2023-12-01 to 2024-12-31
  Both systolic and diastolic Blood Pressure levels of enrolled patients
creatinine | 2023-12-01 to 2024-12-31
  creatinine levels of enrolled patients
urea nitrogen | 2023-12-01 to 2024-12-31
  urea nitrogen levels of enrolled patients